CLINICAL TRIAL: NCT01480505
Title: Primary Vitrectomy for the Treatment of Retinal Detachment in Highly Myopic
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Nicot Frederic, Docteur, Centre Hospitalier Universitaire Dijon
Other Study IDs: Brice 01
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Intraocular Pressure,; Postoperative Complications
Keywords: Retinal detachment; high myopia; macular hole; axial length; Scleral buckling; Vitrectomy; Visual acuity; fundus examination results
MeSH Terms: conditions — Postoperative Complications; Retinal Detachment; Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High myopic eye: Persons with high Myopia suffered from Rhegmatogenous Retinal detachment
  Interventions: Procedure: Pars plana vitrectomy with gas tamponade

INTERVENTIONS:
Procedure: Pars plana vitrectomy with gas tamponade — A standard three-port 20 Gauge vitrectomy under a wide-angle-viewing contact lens was performed. Peripheral vitreous shaving was completed under slit-lamp illumination without contact lens by gentle scleral indentation. Posterior hyaloid detachment was checked and completed if necessary without dye. The epiretinal membrane removal or internal limiting membrane (ILM) peeling was performed if necessary. In general this latter procedure was not conducted for RD secondary to peripheral retinal tears without any sign of PVR or ERM but was done in almost all cases related to posterior break.
  Subretinal fluid was aspirated through the retinal tear, the MH, the PVT or through a retinotomy to obtain a complete peroperative retinal reattachment.

SUMMARY:
Purpose:

To assess the functional and anatomical outcome of primary vitrectomy without scleral buckling for rhegmatogenous retinal detachment (RRD) in highly myopic eyes with axial length over 30 mm.

Methods Design: Retrospective single center series. Setting: University Hospital. Patients: High myopic patients treated with primary vitrectomy without scleral buckling for a rhegmatogenous retinal detachment.

Outcome measures: Anatomical success rate with complete reattachment of the retina without silicone oil tamponade and postoperative best-corrected visual acuity (BCVA).

ELIGIBILITY:
Inclusion Criteria:

* retinal detachment secondary to peripheral breaks (retinal tears, atrophic retinal hole)
* secondary to posterior breaks (MH, PVT).

Exclusion Criteria: retinal detachment secondary to

* severe eye injury,
* diabetic retinopathy,
* retinopathy of prematurity,
* uveitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On the basis of axial length greater than 30 mm, 67 eyes of 67 patients with at least six-month follow-up in our department were selected.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 1999-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Assessing the functional and anatomical outcome of primary vitrectomy in Rhegmatogenous retinal detachment in highly myopic eyes
  To assess by visual acuity measurements, fundus ophthalmoscopy and OCT scans the functional and anatomical outcome in patients with higly myopic eyes whom we performed primary vitrectomy without scleral buckling for rhegmatogenous retinal detachment (RRD)in comparison to standard surgical technics wich consist on scleral buckling and pars plana vitrectomy with fluid gas exchange.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department, Dijon, Burgundy, France